CLINICAL TRIAL: NCT06454695
Title: Improving Treatment of Severe Major Depressive Disorder by Reducing Negative Future-Oriented Mental Imagery
Brief Title: Improving Treatment of Major Depressive Disorder by Reducing Negative Future-Oriented Mental Imagery
Acronym: PROFIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: GGZ Eindhoven (participating site) (Unknown); Mental Care Group (i.e., HSK group and Mentaal Beter; participating sites) (Unknown); Praktijk V (participating site) (Unknown); ZonMw (funding) (Unknown); Depressie Vereniging (patient association) (Unknown); MIND (civil society organization) (Unknown)
Responsible Party: Principal Investigator, Claudi Bockting, Prof dr Claudi Bockting, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2023.0973; NL85551.018.23 (Other: ToetsingOnline)
Record Dates: First submitted 2024-05-23; First posted 2024-06-12 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Major Depressive Disorder; Mental Imagery; Cognitive Behavioral Therapy
Keywords: Imagery rescripting; Prospective negative mental images; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: The design is a randomized, controlled, pragmatic, multicenter, pilot trial. Adult patients with major depressive disorder will be randomized (1:1) to either treatment as usual (TAU) only, or TAU with future-oriented imagery rescripting.
Who Masked: Outcomes Assessor
Masking Description: Most questionnaires will be self-reported via Castor EDC. Only a screening interview will be administered by researchers online.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (Active Comparator): Participants receive Treatment as Usual (TAU) for their depression (i.e., psychotherapy and/or medication).
  Interventions: Other: Treatment as Usual
- Imagery Rescripting (Experimental): Participants receive Treatment as Usual (TAU) for their depression (i.e., psychotherapy and/or medication) plus 3-5 future-oriented imagery rescripting therapy (45 minutes weekly sessions).
  Interventions: Behavioral: Future-oriented imagery rescripting; Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Future-oriented imagery rescripting — In this pilot study, in the screening phase, negative or catastrophic future-oriented images will be explored for all patients, including ratings of distress. The future-oriented imagery rescripting consists of 3-5 sessions; each image will be treated in one session, starting with the image that causes highest distress. The protocol is largely based on Hackmann (1998), with minor adaptations from other protocols.
  Arms: Imagery Rescripting
Other: Treatment as Usual — Psychotherapy and/or medication

SUMMARY:
Patients with major depressive disorder (MDD) often do not sufficiently benefit from treatment. That is, around 50% of patients with MDD do not respond to treatment and 20-30% only achieve partial remission. Future-oriented negative mental imagery (e.g., mental images of suicide or own funeral) is likely an important maintaining factor of depression and initial studies in depression indicate that targeting mental imagery with 'imagery rescripting' could be a promising therapeutic technique to reduces depressive symptomatology by targeting these images directly that elicits strong affects/emotions and depressive symptomatology.

Before testing the (cost)effectiveness of future-oriented imagery rescripting to treatment as usual (TAU), a pilot study is needed to examine 1) the acceptability of the intervention, 2) the feasibility of the study, and 3) the variance of effect on reducing depressive symptomatology that can serve as estimate of the sample size for a follow-up randomized controlled trial (RCT).

A multicenter pilot RCT with a mixed factorial design with three time points (i.e., baseline, post-treatment, and follow-up of 3 months) will test 50 patients with MDD who will be randomly allocated to future-oriented imagery rescripting plus TAU or TAU only.

The sample consists of adult patients of 18 years or older with an MDD diagnosis.

All patients in this pilot study receive TAU, which involves a combination of pharmacological and psychological interventions. Half of the patients will also receive 3-5 sessions of future-oriented imagery rescripting (ImRes). In each ImRes session, patients identify an image of a autobiographic catastrophic future event (e.g., catastrophic images of future suicide or the loss of work or a loved one). They are subsequently asked to "rescript" this image into a more benign one.

The primary aim of this pilot study is to determine the acceptability of the intervention. The secondary aims are to elucidate factors that may facilitate or hinder the feasibility of the follow-up RCT (e.g., recruitment process) and to estimate the variance of the effect on reduction of depressive symptomatology, which informs the sample size calculation of the follow-up RCT. To study acceptability, the investigators assess depressive symptoms (BDI-II and BADS) and treatment satisfaction (SRS and CSQ-8). To measure feasibility, the investigators will assess recruitment/admission ratio, dropout and (serious) adverse events. Finally, to estimate the variance of effects, group effects on the BDI-II will be tested at post-treatment and follow-up (corrected for baseline).

Imagery rescripting on negative memories has already proven effective and safe in MDD patients. There is no known major risk associated with study participation. Patient burden comprises an online or phone-based screening interview of maximum 60 minutes and several questionnaires. Participants receive a reimbursement of €25,- after study completion (i.e., after follow-up assessment). The project will contribute to improving the care for patients with MDD. If the results show that the intervention is feasible and acceptable, this pilot study will inform the setup of the main RCT on the (cost)effectiveness of the intervention (ZonMW).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older;
* Meet DSM-5 criteria for major depressive disorder;
* Presence of 1-3 negative future-oriented mental images, which cause distress;
* Be able to understand questionnaires and study information letter;
* In case of medication use: are stable on medication for six weeks or longer.

Exclusion Criteria:

* Current or history of psychotic disorder;
* Current or history of bipolar disorder;
* Severe cognitive impairment (e.g., mental retardation) as evidenced by educational records, parental report and/or clinical impression;
* Current EMDR or imagery rescripting therapy;
* Other circumstances that might affect participation (e.g., severe medical disorder, relocation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory (Acceptability) | From baseline to the end of the study at follow-up (total of 18 weeks).
  Beck Depression Inventory (BDI-II) for depressive symptoms, consisting of 21 questions with scores between 0-3 whereby a higher score indicates a worse outcome.
Behavioral Activation for Depression Scale (Acceptability) | From baseline to the end of the study at follow-up (total of 18 weeks).
  Behavioral Activation for Depression Scale (BADS-NL) for depressive symptoms, consisting of 25 questions with scores between 0-6 whereby a higher score indicates a worse outcome.
Session Rating Scale (Treatment satisfaction) | During treatment intervention (total of 5 weeks)
  Session Rating Scale (SRS) is filled in during the intervention, consisting of 4 visual analogue scales ranging between 0-100.
Client satisfaction Questionnaire (treatment satisfaction) | After the study intervention and at follow-up
  Client Satisfaction Questionnaire (CSQ-8), consisting of 8 questions whereby the answers ranged from totally disagree to totally agree

SECONDARY OUTCOMES:
Recruitment/admission ratio (Feasibility) | From enrollment to the end of the study at follow-up (total of 18 weeks).
  Recruitment/admission ratio.
Dropout (Feasibility) | From enrollment to the end of the study at follow-up (total of 18 weeks).
  Dropout.
(serious) adverse events (Feasibility) | From enrollment to the end of the study at follow-up (total of 18 weeks).
  (serious) adverse events.
Variance of effect | From enrollment to the end of the study at follow-up (total of 18 weeks).
  Group effects on the Beck Depression Inventory (BDI-II) will be tested at post-treatment and 3 months follow-up (corrected for baseline).

OTHER OUTCOMES:
Structured Clinical Interview for DSM-5 | Screening
  Structured Clinical Interview for DSM-5; SCID-5 - Dutch version: sections on depressive disorders, psychotic disorder, anxiety disorders, substance use disorder and posttraumatic stress disorder
Positive and Negative Affect Schedule | From baseline to the end of the study at follow-up (total of 18 weeks).
  Positive and Negative Affect Schedule (PANAS) for affect, consisting of 20 questions with scores between 1-5. For the total positive score, a higher score indicates more of a positive affect. For the total negative score, a lower score indicates less of a negative affect.
5-level EQ-5D | From baseline to the end of the study at follow-up (total of 18 weeks).
  5-level EQ-5D (EQ-5D-5L) for quality of life, consisting of 5 questions with scores between 1-5 whereby a higher score indicates a worse outcome.
Generalized Anxiety Disorder | From baseline to the end of the study at follow-up (total of 18 weeks).
  Generalized Anxiety Disorder questionnaire (GAD-7) for anxiety, consisting of 7 questions with scores between 0-3 whereby a higher score indicates a higher burden.
Rating of mental images | From baseline to the end of the study at follow-up (total of 18 weeks).
  Rating of mental images on emotions, vividness, uncontrollability, distress and core belief, using a visual analogue scale, ranging from 0-100 whereby a higher score indicates a high level of presence.
Prospective Imagery Task | From baseline to the end of the study at follow-up (total of 18 weeks).
  Prospective imagery task (PIT) for vivedness and likelihood of mental images, consisting of 20 questions with scores between 0-5, whereby a higher score indicates a higher possibility.
Monitoring of Treatment as Usual | From baseline to the end of the study at follow-up (total of 18 weeks).
  Monitoring of 'Treatment as Usual' (TAU) via their therapist. "Which therapy has the patient received (including medication + dose; possible in-patient treatment)?"

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC (location AMC), Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
Very sensitive information.